CLINICAL TRIAL: NCT04105582
Title: Phase I Clinical Study of Immunotherapy With Personalized Synthetic Vaccines in Patients With Triple Negative Breast Cancer
Brief Title: Breast Cancer Neoantigen Vaccination With Autologous Dendritic Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: Fundación Salud de los Andes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TEBICA002
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: Dendritic cells; Neo-antigen; Personalized medicine; immunotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neo-antigen pulsed Dendritic cell (Experimental): Autologous dendritic cells pulsed with tumor-specific neo-antigen (synthetic peptide)
  Interventions: Biological: Neo-antigen pulsed Dendritic cell

INTERVENTIONS:
Biological: Neo-antigen pulsed Dendritic cell — Patients that have already finished their conventional treatment (chemotherapy and/or surgery) will be vaccinated with dendritic cells pulsed with synthetic peptide

SUMMARY:
In this project, the investigators propose the first clinical study in Colombia of vaccination of patients with triple-negative breast cancer (TNBC) using synthetic peptides that contain mutations of the tumor itself that will be presented to the immune system by autologous dendritic cells to assess immunogenicity and safety of this type of personalized vaccine. Achieving the specific objectives set out in this project will mean that the investigators can validate in Colombia the experimental design necessary to identify exclusive epitopes in the tumors of the participants in this study, and also that have been able to demonstrate the safety and immunogenicity of these vaccines.

DETAILED DESCRIPTION:
EXECUTIVE SUMMARY.

The achievements of personalized medicine in cancer research in developed countries make envision that various types of cancer in an advanced stage, will be in the medium term treatable diseases. The discovery of new therapies is the product of the achieved development of Translational Medicine (the laboratory findings translated in short term to the patient benefits), a new approach to applied medicine led by researchers in the universities in alliance with the private sector who carry out clinical studies. Despite the advances of Personalized and Translational Medicine in the developed world in Colombia, this discipline has an incipient development.

Due to its genetic instability, triple-negative breast cancer - (CMTN) (ER-, PR-, Her2 / neu-) among other tumors with a high number of mutations makes it resistant to chemotherapy/radiotherapy regimens generating high morbidity and mortality. Furthermore, genetic instability contributes not only to the immuno-editing of these tumors [5] but to the generation of a suppressive tumor microenvironment [6], which are factors that contribute to the escape of these tumors to their immunosurveillance [7, 8]. However, recent achievements suggest that these factors are controllable using personalized medicine. While immunosuppression is modulated with the use of anti-checkpoint antibodies ("anti-check points" such as anti-CTLA4, anti-PD1, and anti-PDL-1) [9], genetic instability that generates tumor neoantigens, may become the Achilles' heel of these tumors. Phase I clinical studies of patients with melanoma and lung cancer metastatic treated with Ipilimumab (anti-CTLA4 of anti-PD1) - to decrease immunosuppression - using together with vaccines peptides corresponding to tumor mutations that are presented in MHCI and MHCII molecules and are recognized by LT-CD8 as foreign antigens, led these cells to destroy the tumor efficiently when used as a vaccine [10-13]. For this reason, the identification of non-synonymous mutations of single amino acid and vaccination with 25 amino acid peptides incorporating these mutations (synthetic vaccines), is emerging as an alternative for cancer immunotherapy [10-13] in what is called neoantigen based synthetic cancer vaccines. In an approach that takes 16 weeks, today it is possible to go from the analysis of the tumor transcriptome to identify the universe of tumor mutations up to the vaccination of the patient with peptides containing tumor mutations, with the important clinical response to the tumor not achieved so far in patients with melanoma and non-small cell carcinoma of the metastatic lung [10-13]. Therefore, we propose to carry out the first clinical study in Colombia of vaccination of patients with CMTN using synthetic peptides that contain mutations of the tumor itself that will be presented by autologous dendritic cells in order to evaluate the immunogenicity and safety of this type of personalized vaccine. Achieving the specific objectives set out in this project will mean that we have validated in Colombia the experimental design necessary to identify unique epitopes in each tumor of the participants in the study in addition to demonstrating the safety and immunogenicity of these vaccines. Once this has been achieved, we consider having taken an important step towards implementation in our country of the use of this type of vaccine for immunotherapy not only of CMTN but of other highly fatal tumors such as glioblastoma, gastric, esophagus, and pancreas.

This project is carried out by the National University, the Hospital El Tunal de Bogotá, and the Fundación Salud de los Andes, has the collaboration of Professor Luis Fernando Niño and Andrés Pinzón, experts in bioinformatics in the Universidad Nacional; Dr. Chris Miller at Washington University at the McDonnell Genomic Institute at Washington University, School of Medicine in Saint Louis; has the advice of Dr. Pedro Romero from the University of Lausanne (Switzerland) who has extensive experience in immunotherapy clinical trials of melanoma patients with synthetic peptides as a vaccine and with researchers from the Research Group in Immunology and Clinical Oncology (GIIOC) of the Fundación Salud de los Andes.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient who is prescribed as a treatment for her cancer initiating neo-adjuvant chemotherapy with Doxorubicin / cyclophosphamide (A / C) administered prior to cycles with Taxanes and followed by surgery to remove the tumor.
* Be between 18 and 75 years old.
* That the patient agrees to participate in the Clinical Study prior to the start of chemotherapy.
* Have free venous access.
* Signature of informed consent.

Exclusion Criteria:

* Heart disease.
* Diabetes
* Renal impairment
* Coagulation disorders
* Have been hospitalized in the last month
* Have another active tumor with the exception of skin tumors of the squamous-cell or basal-cell carcinoma.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Adverse effects and Safety | One year after innoculation
  Number of participants with a treatment-related adverse event as associated with dendritic cells and neo-antigen inoculation assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Neoantigen Immunogenicity | 6 months after last innoculation
  Measurement of T cell response against tumor-specific neo-antigen assessed by interferon gamma release by ELISPOT or ELISA of in vitro culture of T cells and mutated peptide-pulsed dendritic cells, normalized against wild type peptide.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Parra-Lopez, MD PhD, Principal Investigator — Full Professor School of Medicine. Microbiology Department.
Locations (1):
- Universidad Nacional de Colombia, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No
We are not going to share individual participant data (IPD)